CLINICAL TRIAL: NCT06700811
Title: Phase 1 Study of Ketogenic Diet for Prevention of Epileptic Spasms in Infantile Onset Genetic Epilepsies
Brief Title: Ketogenic Diet for Prevention of Epileptic Spasms in Infantile Onset Genetic Epilepsies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Heather Olson (Other)
Collaborators: Boston Children's Hospital Translational Research Program (TRP) Pappendick Family Therapeutic Acceleration Award (Unknown)
Responsible Party: Sponsor-Investigator, Heather Olson, Assocaite Professor of Neurology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P00047586
Record Dates: First submitted 2024-11-12; First posted 2024-11-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Developmental and Epileptic Encephalopathies; Epileptic Spasms; Genetic Epilepsy; Neonatal and Infant Epilepsy
Keywords: Ketogenic diet; Epileptic spasms prevention; epilepsy; infantile spasms; epileptic spasms; seizures; infant; eeg; open label; Phase 1; dietary treatments; developmental and epileptic encephalopathy; genetic; prevention; epileptic encephalopathy; refractory epilepsy
MeSH Terms: conditions — Spasms, Infantile; Epilepsy; Seizures; Drug Resistant Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: All subjects will receive treatment with ketogenic diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet (Experimental): KetoVie® 4:1 Formula will be administered by oral feeding or gastrostomy tube as indicated. The duration of the diet will be from the time of enrollment up to 12 months of age or until 3 months after a diagnosis of Epileptic Spasms (range 3-15 months).
  Interventions: Drug: Ketogenic diet

INTERVENTIONS:
Drug: Ketogenic diet — The ketogenic diet formula will be KetoVie®, supplied by Ajinomoto Cambrooke. Ketogenic diet ratio will aim to achieve ketosis, with a minimum level of beta-hydroxybutyrate of 1.0mmol/L. Ratios of ketogenic diet generally range from 1:1 to 4:1. Ratio will increase per standard clinical care for ketogenic diet initiation. For the trial we will aim to reach a maximum of 4:1 by the 6 week follow-up visit, but stopping at a lower ratio if BHB is ≥ 5mmol/L, CO2 ≤ 18 mmol/L, for tolerance, or to meet protein needs. A minimum 1:1 ratio is required to continue in the trial. Ratios higher than 1:1 are often required to obtain ketosis of ideally 2-5mmol/L in infants.

SUMMARY:
Epileptic spasms (ES) are a predominantly infantile seizure type observed frequently in certain genetic disorders. Ketogenic diet (high ratio of fat to carbohydrate/protein) is an established non-medication treatment for difficult to control seizures, including ES. Because ES are associated with worse developmental and cognitive outcomes if not detected or treated quickly and effectively, this trial aims to test the ketogenic diet to prevent ES in this high-risk population. This trial is a single-center pilot study of 10 infants with genetic seizure disorders to establish if the protocol of early ketogenic diet administration and ES evaluation is safe and feasible.

DETAILED DESCRIPTION:
Epileptic spasms (ES) are a highly prevalent and often refractory form of seizures in genetic Developmental and Epileptic Encephalopathies (DEEs), affecting 55% of patients. Prevalence is higher in subsets such as CDKL5 Deficiency Disorder (82%). Infantile epileptic spasms syndrome can be associated with developmental regression, and early and effective treatment of ES impacts developmental outcomes. Diagnosis of ES, made by a combination of clinical history and EEG, can be delayed if ES are subtle or mixed with other seizure patterns. Clinical experience and the literature support use of the ketogenic diet for refractory epilepsy in infancy, including ES, particularly for some established genetic diagnoses. Further, there is precedent for preventing seizures, including ES, in Tuberous Sclerosis Complex with vigabatrin. The hypothesis of this investigation is that treatment of infants with genetic DEEs with the ketogenic diet will prevent the development of ES, or, if ES do develop, improve treatment response to standard therapy. The focused goal of this proposal is to demonstrate feasibility of initiating and maintaining ketogenic diet in infants with genetic DEEs, with serial EEG monitoring. This trial is a prospective, open-label treatment with ketogenic diet (goal ratio 4:1) in 10 infants with genetic DEE (seizure onset <6 months). The trial will evaluate adherence to ketogenic diet, starting within 6 weeks of enrollment, with a primary endpoint of maintaining a minimum ratio of 1:1 through 3 months after ES onset (12 months of age if they do not develop ES). The trial will evaluate adherence to EEG testing every 6 weeks. This work will lay the foundation for a multi-center Phase 2 trial.

ELIGIBILITY:
Inclusion Criteria:

* Plan for initiation of ketogenic diet by clinical team for treatment of epilepsy
* The clinical team initiating the ketogenic diet agrees that the use of the KetoVie formula is appropriate for the subject, as all study subjects need to receive the same formula
* Male or female, age 0 to less than 9 months (including neonates per investigator's judgment)
* Epilepsy onset at less than 6 months of age
* Abnormal development (any sub score of the Bayley-4 less than 1 standard deviation below the mean) and/or neurologic exam (microcephaly, macrocephaly, strabismus, abnormal vision/CVI, hypotonia, spasticity, dystonia, movement disorder), per investigators judgment
* Genetic epilepsy diagnosis, pathogenic or likely pathogenic variant(s) with consistent phenotype and inheritance pattern
* Weight adequate to complete required study laboratory testing without exceeding maximum allowable blood draws per draw or in a 30 day period per BCH policy

Exclusion Criteria:

* Epileptic spams prior to enrollment
* Tuberous sclerosis complex, trisomy 21 (based on differential response to ES treatment)
* Metabolic diagnosis with targeted treatment (including specific indication for ketogenic diet such as glucose transporter disorder, vitamin dependent epilepsies, and others) or exclusion for the ketogenic diet
* Ongoing treatment with vigabatrin, ACTH, corticosteroids, topiramate or zonisamide. Other anti-seizure medications are permitted.

Ages: 0 Days to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Achievement of ketosis | rom ketogenic diet initiation until 3 months after the diagnosis of ES (if it occurs) or until 12 months of age
  Proportion of subjects assigned to ketogenic diet who achieve ketosis by 6 weeks and maintain a minimum ratio of 1:1 through 3 months after onset of epileptic spasms (ES) or 12 months of age
EEG compliance | From ketogenic diet initiation until the onset of ES (if it occurs) or until 12 months of age
  Proportion of subjects who complete EEGs every 6 weeks (+/- 2 weeks) until onset of ES or 12 months of age

SECONDARY OUTCOMES:
Epileptic Spasms Outcome | From ketogenic diet initiation until 12 months of age
  Proportion of subjects who develop ES by 12 months of age
EEG Outcome | From ketogenic diet initiation until 12 months of age
  Proportion of enrolled subjects for whom a study EEG identified ES or identified hypsarrhythmia with subsequent workup leading to diagnosis of ES prior to clinical suspicion
Safety Outcome | From ketogenic diet initiation until the diet is weaned (up to 18 months of age)
  To assess safety of ketogenic diet treatment in infants with genetic DEEs by monitoring the rate of serious adverse events and adverse events, expected and unexpected

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No